CLINICAL TRIAL: NCT04277910
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, SAD/MAD Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MT2004
Brief Title: A SAD/MAD Study to Evaluate the Safety, Tolerability, PK and PD of MT2004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xi'an Biocare Pharma Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT2004-I-A01; NCT04768452 (obsolete NCT alias)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, sequential parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT2004 (Active Comparator): MT2004 oral capsules treated group
  Interventions: Drug: MT2004
- Placebo (Placebo Comparator): Placebo oral capsules treated group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT2004 — MT2004 oral capsules
  Arms: MT2004
Drug: Placebo — Placebo oral capsules
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of a single dose of MT2004 following oral single and multiple ascending dose administration.

DETAILED DESCRIPTION:
A total of 48 subjects will be evaluated with 36 subjects randomized to receive active drug and 12 subjects randomized to receive placebo in a double-blind fashion (eight subjects per each dose cohort, six subjects randomized to active drug and two subjects randomized to placebo). A separate open panel of 8 subjects will receive a single dose of MT2004 under fed conditions following the last of the SAD dose escalation cohorts. The dose level will be selected by the sponsor based upon the safety and PK data generated in each dose escalation cohort of the SAD part of the trial. A total of 24 subjects will receive MT2004 (8 subjects in each dose cohort for a total of 3 cohorts, 6 subjects randomized to active drug and 2 subjects randomized to placebo per cohort). MT2004 dosing regimens (dose levels and duration of administration) will be determined based on the collective SAD PK and safety data from Part 1 and nonclinical data of MT2004 (pharmacology and toxicology). Tentative dosing regimen is once daily for a consecutive 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 55 years, inclusive;
3. Female subjects have a negative urine pregnancy test result at screening and Day -1, and meet one of the following criteria:

   * Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   * Surgically sterile for at least 3 months prior to screening by one of the following means:
   * Bilateral tubal ligation
   * Bilateral salpingectomy (with or without oophorectomy)
   * Surgical hysterectomy
   * Bilateral oophorectomy (with or without hysterectomy)
   * Postmenopausal, defined as the following:
   * Last menstrual period greater than 12 months prior to screening
   * Postmenopausal status confirmed by serum follicle stimulating hormone (FSH) and estradiol levels at screening;
4. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12- lead ECG, and vital signs;
5. Normal renal function as determined by Investigator following review of clinical laboratory test results;
6. Non-smoker and no more than 2 tobacco-containing products including nicotine replacement products in last 6 months;
7. Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive and body weight not less than 50 kg;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center.
9. Male subjects with female partners of child bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Known or suspected malignancy;
3. History of pancreatitis or gall stones;
4. History of unexplained syncope, symptomatic hypotension or hypoglycemia;
5. Family history of long QTc syndrome;
6. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
7. History of organ transplantation with the exception of cornea transplantation;
8. Poor venous access;
9. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
10. Donated or lost >500ml of blood in the previous 3 months;
11. Taken an investigational drug or participated in a clinical trial within 3 months (or 5 half- lives), whichever is longer;
12. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the first dose of study drug;
13. Hospital admission or major surgery within 6 months prior to screening;
14. A history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
15. A history of alcohol abuse according to medical history within 9 months prior to screening;
16. A positive screen for alcohol and/or drugs of abuse at screening or Day

    -1;
17. An unwillingness or inability to comply with food and beverage restrictions during study participation;
18. Use of over-the-counter (OTC) medication within 7 days, and herbal (including St John's Wort, herbal teas, garlic extracts) within 7 days prior to dosing (Note: Use of acetaminophen at < 2 g/day is permitted until 24 hours prior to dosing);
19. Pregnant or breast feeding at screening or planning to become pregnant during the study;
20. Inability to swallow multiple capsules simultaneously
21. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Cmax of MT2004 | 48 hours
  Maximum observed concentration (Cmax) of MT2004
AUClast of MT2004 | 48 hours
  Area under the concentration-time curve (AUC) from Hour 0 to the last measurable concentration (AUC0-last) of MT2004
Tmax of MT2004 | 48 hours
  Time to maximum concentration (Tmax)
T half of MT2004 | 48 hours
  T half of MT2004
Plasma FGF19 Level | 24 hours
  Plasma FGF19 Level
Serum 7-alpha-hydroxy-4-cholesten-3-one (C4) Level | 24 hours
  Serum 7-alpha-hydroxy-4-cholesten-3-one (C4) Level

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator — Pharmaron CPC, Inc.
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No